CLINICAL TRIAL: NCT03648047
Title: Efficacy of a Digital Kinematic Biofeedback System for Rehabilitation After Arthroscopic Rotator Cuff Repair Versus Conventional In-person Rehabilitation: a Randomized Controlled Study
Brief Title: Digital Biofeedback System Versus Conventional Rehabilitation After Rotator Cuff Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic imposed restrictions to normal study conduct
Sponsor: Sword Health, SA (Industry)
Collaborators: Hospital da Prelada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH-RCT-ARCR-01
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All patients will be assessed by an independent outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in this group will receive a mixed home-based rehabilitation program consisting of face-to-face sessions with a Physical Therapist (with decreasing periodicity depending on program stage) as well as sessions performed with a digital kinematic biofeedback system.
  Interventions: Device: Digital kinematic biofeedback device; Other: Additional face-to-face rehabilitation sessions
- Conventional rehabilitation (Active Comparator): Patients in this group will receive a home-based rehabilitation program consisting of face-to-face sessions with a Physical Therapist 3 times per week, for 1 hour. Patients will also be instructed to perform additional unsupervised sessions in at least two other days of the week. Compliance to these additional sessions is not mandatory, but patients will be asked to fill in a diary regarding these extra-sessions.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Digital kinematic biofeedback device — The system will be used independently by the patients to perform rehabilitation sessions at home, under remote monitoring from the clinical team.
  Other Names: SWORD Phoenix
  Arms: Experimental group
Other: Conventional rehabilitation — Patients will receive conventional face-to-face sessions by a Physical Therapist.
  Arms: Conventional rehabilitation
Other: Additional face-to-face rehabilitation sessions — Patients will receive face-to-face sessions in addition to sessions performed with the Digital Rehabilitation Device
  Arms: Experimental group

SUMMARY:
This study was designed to compare the clinical outcomes of a mixed home-based rehabilitation program after arthroscopic rotator cuff repair, incorporating face-to-face sessions as well as sessions performed with a novel digital kinematic biofeedback system against conventional in-person home-based rehabilitation, with the intent of reducing the need for face-to-face sessions.

The investigators hypothesize that the clinical outcomes of such a program will be at least similar to those of conventional rehabilitation.

Patients will be enrolled pre-operatively and then randomized into 2 groups: experimental group and conventional rehabilitation group. Both groups will perform a 12 to 16-week rehabilitation program starting immediately after surgery.

Outcomes will be measured at baseline, 8 and 12 weeks. In patients where a decision is made to extend the program to 16 weeks, another assessment will be made at this point.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain and functional limitation with clinical examination compatible with rotator cuff tendinopathy
* Imaging (MRI or ultrasound) evidence of rotator cuff tear (supra and/or infraspinatus tendon tear inferior to 3 cm? or 5cm?)
* Indication for a simple rotator cuff repair according to the patient´s orthopedic surgeon
* Ability to understand simple and complex motor commands
* Availability of a carer to assist the patient after surgery

Exclusion Criteria:

* Patients admitted for revision cuff repair
* Complex cuff tears (involving subscapularis tendon or more than one tendon besides supra and infraspinatus, or massive dimension tears)
* Glenohumeral arthritis
* Irreparable tendon defect
* Patients with concomitant neurological disorders (ex. Stroke, Parkinson´s disease, multiple sclerosis)
* Aphasia, dementia or psychiatric comorbidity interfering with the communication or compliance to the rehabilitation process
* Respiratory, cardiac, metabolic conditions or others incompatible with at least 30 minutes of light to moderate physical activity
* Major medical complications occurring after surgery that prevent the discharge of the patient within 10 days after surgery
* Other medical and/or surgical complications that prevent the patient from complying with a rehabilitation program
* Blind and/or illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Constant Score Test | Baseline, 8 weeks after surgery, 12 (and 16) weeks.
  The Constant Score is a functional assessment score specific to the shoulder region. It is the most used instrument to assess the shoulder in Europe and its psychometric properties prove it to be a valid, reliable and responsive measure.

SECONDARY OUTCOMES:
Change in QuickDASH score | Baseline, 8 weeks after surgery, 12 (and16) weeks.
  The QuickDASH is an 11-item self-administered outcome measure, specific to measure disability and symptoms in individuals with musculoskeletal disorders of the upper limb.It is an instrument widely used for clinical or research purposes and which has proven to be a valid, reliable and responsive measure.
Change in Shoulder Range of Motion | Baseline, 8 weeks after surgery, 12 (and16) weeks.
  Shoulder range of motion (in degrees) in the following exercises: sitting external rotation/abduction/flexion; lying internal/external rotation with 90º shoulder abduction

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — SWORD Health; Rosmaninho Seabra, MD, Study Chair — Hospital da Prelada
Locations (1):
- Hospital da Prelada, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon study publication, for 5 years.
Access Criteria: Study protocol will be available through a direct link in this platform. The excel file with the aggregate results will be made available as supplementary information upon study publication.
URL: https://drive.google.com/file/d/1BBfowtHXm4U91QTRPilzvxOFglKx3T_h/view?usp=sharing

REFERENCES:
- [Derived] Correia FD, Molinos M, Luis S, Carvalho D, Carvalho C, Costa P, Seabra R, Francisco G, Bento V, Lains J. Digitally Assisted Versus Conventional Home-Based Rehabilitation After Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Mar 1;101(3):237-249. doi: 10.1097/PHM.0000000000001780. PMID 33935152

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03648047/Prot_SAP_000.pdf